CLINICAL TRIAL: NCT05688644
Title: Efficacy and Safety of Sacral Neuromodulation With InterStim II in Neurogenic Bladder and/or Bowel Patients
Brief Title: Sacral Neuromodulation in Neurogenic Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Omri Schwarztuch Gildor (Other)
Responsible Party: Sponsor-Investigator, Omri Schwarztuch Gildor, Urologist, Clalit Health Services
Organization: Clalit Health Services (Other)
Other Study IDs: MMC-0221-21
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Neurogenic Bladder; Neurogenic Bowel; Urge Incontinence; Overactive Bladder; Retention, Urinary; Fecal Incontinence
Keywords: Sacral Neuromodulation; Neurogenic Bladder; Neurogenic Bowel
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Neurogenic Bowel; Urinary Incontinence, Urge; Urinary Bladder, Overactive; Urinary Retention; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Neurogenic Patients: Patients with underlined relevant neurologic condition, with either neurogenic bladder or bowel, after advanced evaluation of InterStim II
  Interventions: Device: InterStim II
- Idiopathic: Patients without underlined relevant neurologic condition, after advanced evaluation of InterStim II
  Interventions: Device: InterStim II

INTERVENTIONS:
Device: InterStim II — Sacral neuromodulation

SUMMARY:
The goal of this observational study is to evaluate efficacy and safety of sacral neuromodulation in neurogenic patients compared to non-neurogenic (idiopathic) patients. [. The main question[s] it aims to answer are:

* determine efficacy and safety of the therapy in neurogenic patients.
* compare outcomes of the therapy to idiopathic patients.

If there is a comparison group: Researchers will compare the outcomes of the therapy between the neurogenic and non-neurogenic subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent InterStim II advanced evaluation for approved indication

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with approved indication for sacral neuromodulation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Decrease of at least 50% in number of catheterizations per day | 1 year
Decrease of at least 50% in number of fecal incontinence episodes | 1 year
Decrease of at least 50% in number of urge urinary incontinence episodes | 1 year

SECONDARY OUTCOMES:
Number of revision surgeries | 1 year
number of follow-up visits for programming and/or troubleshooting | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No